CLINICAL TRIAL: NCT03560804
Title: Use of Impedance Cardiography and Applanation Tonometry for Prediction of the Antihypertensive Effect. Comparison Between an ATII Receptor Antagonist and a Diuretic.
Brief Title: Use of Impedance Cardiography and Applanation Tonometry for Prediction of the Antihypertensive Effect of Two Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHEPA University Hospital (Other)
Responsible Party: Principal Investigator, Maria Pikilidou, MD, MSc, PhD, Post-doctoral researcher, AHEPA University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100
Record Dates: First submitted 2015-01-15; First posted 2018-06-18 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Arterial Stiffness; Ambulatory Blood Pressure Monitoring
Keywords: olmesartan; chlorthalidone; hemodynamics
MeSH Terms: interventions — olmesartan; Chlorthalidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olmesartan (Active Comparator): ARB administration (OLMESARTAN) at a starting dose and titrating at 15 weeks according to reach blood pressure target
  Interventions: Drug: Olmesartan
- Chlorthalidone (Active Comparator): Diuretic administration (chlorthalidone) at a starting dose and titrating at 15 weeks according to reach blood pressure target
  Interventions: Drug: Chlorthalidone

INTERVENTIONS:
Drug: Olmesartan — Administration of olmesartan at starting dose and titrating in order to reach the target blood pressure.
  Other Names: Olartan
  Arms: Olmesartan
Drug: Chlorthalidone — Administration of chlorthalidone at starting dose and titrating in order to reach the target blood pressure.
  Other Names: Hygroton
  Arms: Chlorthalidone

SUMMARY:
The principal aim of the study is to determine whether the hemodynamic parameters measured with the two methods -impedance cardiography and applanation tonometry- can be predictive of the antihypertensive effect of two different classes of drugs, ATII antagonists and diuretics.

The drugs that will be used in the study are olmesartan and chlorthalidone and the duration of the study is 12 months.

The other basic aim of the study is to determine whether there is a difference (>6mmHg) between the two drugs regarding the reduction of the mean 24hour blood pressure and the effect of them on the hemodynamic parameters.

The hemodynamic parameters that will be measured by applanation tonometry are augmentation index, central blood pressure and pulse wave velocity.

The hemodynamic parameters that will be measured by impedance cardiography are cardiac index, thoracic fluid content index, systemic vascular resistance index and others.

DETAILED DESCRIPTION:
The principal aim of the study is to determine whether the hemodynamic parameters measured with the two methods -impedance cardiography and applanation tonometry- can be predictive of the antihypertensive effect of two different classes of drugs, ATII antagonists and diuretics.

The drugs that will be used in the study are olmesartan and chlorthalidone and the duration of the study is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Drug naive patients with 1st or 2nd grade Arterial Hypertension according to the ESH/ESC guidelines 2013
* The patient has signed the concent form

Exclusion Criteria:

* Secondary Hypertension
* 3rd grade of Arterial Hypertension
* Chronic renal failure
* Diabetes Mellitus
* Sleep apnea syndrome
* Chronic or acute inflammatory diseases
* Stroke, myocardial infarction, angina pectoris in the past 6 months
* Heart failure
* Liver disease
* Neoplasms
* Pregnancy
* Valvular Heart disease
* Heigt < 120cm or > 230cm, Weight <30kg or >155kg
* Heart Arrhytmias
* Artificial cardiac pacemaker
* Hemodymanic unstable patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-11-10 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Pulse wave velocity | 12 weeks
  Measured by Sphygmocor devive

SECONDARY OUTCOMES:
Systemic vascular resistance | 12 months
  Measured by impendance cardiography
Ambulatory blood pressure | 12 months
  Daytime and nighttime systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Zebekakis Pantelis, Professor, Principal Investigator — Hypertension Excellence Center, 1st Department of Internal Medicine, AHEPA University Hospital
Locations (1):
- Hypertension Excellence Center, AHEPA University Hospital, Thessaloniki, Greece